CLINICAL TRIAL: NCT04926714
Title: Ophthalmologic Evaluation of Patients With Obesity and Metabolic Syndrome Before and After Bariatric Surgery:A Pilot, Monocentric, Prospective, Open-label Study
Brief Title: Ophthalmologic Evaluation of Patients With Obesity and Metabolic Syndrome Before and After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: XiaoYong Liu (Other)
Responsible Party: Sponsor-Investigator, XiaoYong Liu, Deputy chief physician of opthalmology, The First Affiliated Hospital of Jinan University, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Other Study IDs: 2021JiNanU
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Eye Diseases; Obesity Associated Disorder
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study was to investigate the pathogenic role of obesity on blinding eye diseases in a population of severely obese patients with no history of eye diseases, and to verify whether weight loss induced by bariatric surgery may have a protective effect.

DETAILED DESCRIPTION:
This was a pilot, monocentric, prospective, and open label study conducted at First Affiliated Hospital of Jinan Universityreceived.Patients with body mass index ≥ 32.5Kg/m2; or patients with body mass index of 27.5-32.5Kg/m2 and metabolic diseases were consecutively recruited.All participants underwent complete ophthalmological evaluation， Keratograph 5M and optical coherence tomography.Patients who underwent bariatric surgery were evaluated also 3 months, 6 months and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with BMI≥32.5Kg/m2；
2. patients with BMI27.5-32.5Kg/m2, combined with metabolic diseases;

Exclusion Criteria:

1. Patients with pre-existing ocular diseases or visual alterations were excluded to avoid confounding factors related to pre-existing retinal pathology, independent from obesity per se.
2. Patients with dementia, Parkinson's disease, Alzheimer's disease, multiple sclerosis or other severe neurological diseases were also excluded since ophthalmologic parameters may be altered in these conditions.
3. Patients with lens opacities that made impossible the posterior segment examination, or with a refractive error > +5 or <-8 diopters spherical equivalent were also excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with BMI≥32.5Kg/m2Or patients with BMI27.5-32.5Kg/m2, combined with metabolic diseases;
  2. Subjects understand the purpose of the clinical study and are willing, able and committed to return to the study center for all clinical study visits and to complete all study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
optical coherence tomography | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China